CLINICAL TRIAL: NCT07238621
Title: Evaluation of the Effects of the Serratus Posterior Superior Intercostal Plane Block on Postoperative Pain Levels and Analgesic Requirement in Patients Undergoing Cervical Disc Herniation Surgery
Brief Title: Evaluation of the Postoperative Analgesic Efficacy of SPSIPB in Anterior Cervical Discectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Associate Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2025-07/24
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Anterior Cervical Discectomy; Serratus Posterior Superior Intercostal Plane Block; Postoperative Pain Management; Postoperative Pain; Cervical Disc Herniation
Keywords: postoperative pain; regional anesthesia; opioid free analgesia; ibuprofen; Serratus Posterior Superior Intercostal Plane Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group without peripheral nerve block (Active Comparator): After the patients are monitored, they will be operated under general anesthesia without peripheral nerve block and intraoperative intravenous analgesics (dexketoprofen 50 mg, paracetamol) will be given.
  Interventions: Procedure: Group without peripheral nerve block
- Serratus posterior superior intercostal plane block (Active Comparator): In this study, the intervention will be the SPSIPB. The block will be performed with the patient in the lateral decubitus position.A high-frequency (7-12 MHz) linear transducer will be placed in the transverse plane at the level of the spina scapulae, and the superior medial border of the scapula, the trapezius muscle, the rhomboid muscle, the serratus posterior superior muscle (SPSM), and the second and third ribs will be visualized.
  Subsequently, a sonovisible needle will be advanced just medial to the scapula, targeting the area between the second and third ribs to reach the fascial plane between the SPSM and the intercostal muscles. After the needle makes gentle contact with the rib, 1-2 mL of saline will be used to confirm the correct plane. A total of 30 mL of 0.25% bupivacaine will then be administered into this fascial plane between the SPSM and the intercostal muscle.In the intraoperative period, intravenous analgesics (dexketoprofen 50 mg, paracetamol 1000 mg) will be given.
  Interventions: Procedure: Serratus posterior superior intercostal plane block

INTERVENTIONS:
Procedure: Group without peripheral nerve block — In the postoperative period a ibuprofen dose of 400 mg every 8 hours were administered iv for multimodal analgesia
  Arms: Group without peripheral nerve block
Procedure: Serratus posterior superior intercostal plane block — Serratus posterior superior intercostal plane block will be performed on the patients using 30 ml of 0.25% bupivacaine under ultrasound guidance.Additionally, in the postoperative period a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: Serratus posterior superior intercostal plane block

SUMMARY:
Anterior cervical discectomy is an operation performed for complaints of pain, numbness or loss of strength due to cervical disc disease. With this operation, pressure due to herniation on the upper neck area, spinal cord or nerve roots is relieved. It is performed by microscopic method from the front of the neck.

Nerve blocks reduces opioid consumption in the postoperative period by providing better pain control and therefore has advantages such as fewer side effects and less risk of pulmonary and cardiac complications.

In this study; it was aimed to compare the analgesic effectiveness of serratus posterior superior intercostal plane block and erector spinae plane block, and with the control group in the postoperative period in patients who underwent anterior cervical discectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age who underwent percutaneous nephrolithotomy under general anesthesia and were I-II-III according to the American Society of Anesthesiologists (ASA) risk classification were included in the study.

Exclusion Criteria:

* patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with known allergies to any of the study drugs,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment
* patients who wanted to withdraw from the study,
* patients with alcohol and drug addiction,
* patients with musculoskeletal abnormalitie

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) Scores | Postoperative 24 hours
  Numerical rating scale is used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Total tramadol consumption | Postoperative 24 hours
  Postoperative total analgesic need was recorded as "milligram" in unit.
Quality of Recovery scores | Postoperative 24 hours
  Quality of recovery-15 (QoR15) scale was used for the assessment of patients satisfaction. The scores of QoR15 changes between 0 to 150 points. 0 point means "there is no satisfaction." Higher scores mean indicating a good quality of recovery and better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: ONUR AVCI, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation; ZEYNEP M DEMİRCİ, Study Chair — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation
Locations (1):
- Sivas Cumhuriyet University, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No